CLINICAL TRIAL: NCT02197312
Title: A Clinical Evaluation of NobelProceraTM Bridge Shaded Zirconia
Brief Title: NobelProceraTM Bridge Shaded Zirconia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business reasons
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-159
Record Dates: First submitted 2014-07-03; First posted 2014-07-22 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Posterior Bridge Restoration
Keywords: yttrium-oxide; Y-TZP; bridge; NobelProcera; Shaded Zirconia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NobelProcera Bridge Shaded Zirconia (Other): posterior region
  Interventions: Device: NobelProcera Bridge Shaded Zirconia

INTERVENTIONS:
Device: NobelProcera Bridge Shaded Zirconia

SUMMARY:
Industrial centrally produced 3- or 4-unit bridges of shaded yttrium-oxide partially-stabilized (Y-TZP) zirconia (NobelProceraTM Shaded Zirconia) in combination with a veneering ceramic material will show sufficient CDA ratings and a sufficient survival rate after 5 years

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 (or age of consent), and less than 70 at the time of inclusion.
* The subject is healthy and compliant with good oral hygiene
* The subject is in need of a posterior fixed partial denture restoration 3 or 4 units distal of the canines in the maxilla or mandible.
* The subject shall have a stable occlusal relationship with a fully restored, fixed opposing dentition.
* Obtained informed consent from the subject prior to the study.
* No apical disorder or inflammation of abutment teeth, adjacent and opposing teeth.
* Good gingival / periodontal / periapical status of restoring, opposing and adjacent teeth. Healed situation of soft tissue augmentation is allowed.
* The subject should be available for the 5-year term of the investigation.

Exclusion Criteria:

* The subject is not able to give her/his informed consent to participate.
* Alcohol or drug abuse as noted in patient records or in patient history.
* Reason to believe that the treatment might have a negative effect on the patient's total situation (psychiatric problems), as noted in patient records or in patient history.
* An existing condition where acceptable retention of the restoration is impossible to attain
* Mobility greater than grade 1 of the tooth to be restored.
* Pathologic pocket formation of 4 mm or greater around the tooth to be restored
* Severe bruxism or other destructive habits
* Amount of attached soft tissue is insufficient (attached gingiva less than 2 mm or attachment loss greater than half of the root length).
* Health conditions, which do not permit the restorative procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06-18 (Actual); Primary Completion 2013-11-23 (Actual); Study Completion 2013-11-23 (Actual)

PRIMARY OUTCOMES:
clinical performance of NobelProceraTM Bridge Shaded Zirconia on natural teeth in the posterior region with the proportion of patients with CDA ratings "R" (excellent) or "S"(acceptable) | yearly up to 5 years

SECONDARY OUTCOMES:
survival rate of NobelProceraTM Bridge Shaded Zirconia on natural teeth in the posterior region | yearly up to 5 years

OTHER OUTCOMES:
esthetic performance of NobelProceraTM Bridge Shaded Zirconia on natural teeth in the posterior region as determined by overall patient satisfaction survey | yearly up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Aachen, Aachen, Germany